CLINICAL TRIAL: NCT06525779
Title: Comparison of Requirement of External Laryngeal Manipulation in Double Lumen Tube Insertion With McGrath Laryngoscope vs Macintosh Laryngoscope. A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Principal Investigator, Farah Rasheed, Sanaa Afzal Khan, Shaukat Khanum Memorial Cancer Hospital & Research Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-19-15
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Intubation Complication
Keywords: Double Lumen Tube, External Laryngeal Manipulation, Macintosh, McGrath

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Macintosh Laryngoscope Group (Active Comparator): Patient undergoing intubation with direct laryngoscope using macintosh laryngoscope
  Interventions: Device: Use of macintosh laryngoscope
- McGrath Laryngoscope Group (Active Comparator): Patient undergoing intubation with video laryngoscope using mcGrath laryngoscope
  Interventions: Device: Use of mcGarth laryngoscope

INTERVENTIONS:
Device: Use of macintosh laryngoscope — The requirement of external laryngeal manipulation recorded in use of macintosh vs mcGrath laryngoscope in double lumen tube insertion
  Arms: Macintosh Laryngoscope Group
Device: Use of mcGarth laryngoscope — Use of mcGarth laryngoscope
  Arms: McGrath Laryngoscope Group

SUMMARY:
For anatomical and physiological isolation of the lung, a specialized endotracheal tube known as the double lumen tube (DLT) is used. The introduction of DLT into anesthesia can be attributed to Carlen's who brought forth the concept in 1949. Since then the structure of DLT has continuously evolved. Simplistically speaking; the double lumen tube is a co-axial tube i.e. it contains two tubes put together, the tube with the shorter length stays in the trachea whereas the tube with the longer length enters the right or left main bronchus. If the proximal or tracheal cuff is inflated, air entry is permitted into both lungs. However, if the distal or the bronchial cuff is inflated, ventilation is directed into either lung depending on which lumen has been clamped, at the proximal end of the tube. Conventionally the DLTs were made of red rubber and were reusable but now they have been replaced by disposable plastic tubes which make it easy to view any secretions or blood. Also, since the plastic makes for a thin wall it allows the lumen of the tube to be large enough to allow airflow with minimal resistance. Larger lumens also allow passage of suction catheters and fiber-optic bronchoscope which serves the purpose of confirming correct position of the double lumen tube after placement. Tracheal intubation with a DLT may be facilitated by maneuvers such as external laryngeal manipulation (ELM). It is a simple technique which has been used by anesthetists since many years to enable intubation. Various types of video-laryngoscopes (VL) have been found to perform a crucial part in patients with difficult airways McGrath video-laryngoscope - a portable machine - provides a better laryngeal view compared to Macintosh laryngoscopy, involving cases of intubation involving patients with normal or difficult airways. Though the use of VL for DLT placement has been reported, such studies have fallen short of producing the desired quality of evidence that is required to make a clear determination in favor of one method over the other. It is suggested that more work is needed on this in order to create a wider, more reliable data pool.

DETAILED DESCRIPTION:
After approval from the hospital's institutional review board, a prospective clinical study was conducted at Shaukat Khanum Memorial Cancer Hospital and Research Centre (SKMCH & RC), Lahore, from January 25, 2021 to July 25, 2021. Data was collected from 60 patients that fulfilled the inclusion criteria. Features considered, included patients' demographic including age, gender, co-morbidities and American Society of Anesthesiologist physical status. In addition mallampati score, mouth opening and Wilson score of all patients was recorded as part of routine anesthesia airway assessment. Patients being taken for study were randomly assigned to either of the two groups of 30 each, that is all patients at odd numbers (1, 3, 7, 9 etc.) was allocated to Group 1 (McGrath laryngoscope) whereas all patient at even numbers (2, 6, 8, 10 etc.) was allocated to Group 2 (Macintosh laryngoscope). After explaining the procedure in detail and obtaining an informed consent in the presence of a witness, patients were transferred to the operating room. After standard induction of anesthesia, tracheal intubation using either of the two laryngoscopes depending on group allocation (McGrath laryngoscope or Macintosh laryngoscope) was performed by a designated anesthesia consultant experienced in the use of double-lumen tubes. The requirement of external laryngeal manipulation was recorded on a predesigned checklist.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1, 2, 3 patients
* 18-60 years of age
* Patients undergoing surgery under general anesthesia requiring double lumen tube insertion (e.g. thoracic surgery, three stage esophagectomies)

Exclusion Criteria:

* Patient's refusal
* Patients with cervical spine instability/cervical myelopathy
* Patients requiring rapid sequence intubation
* Patients requiring additional intubation aids like bougie
* Patients having Wilson's Risk Score > 5 (refer to annexure)
* Patients with loose teeth

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
Requirement of External Laryngeal Manipulation | 6 MONTHS
  Requirement of External Laryngeal Manipulation

CONTACTS AND LOCATIONS:
Locations (1):
- Shaukat Khanum Memorial Cancer Hospital and Research Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
no plan yet
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data is available to be shared
Access Criteria: will be available once published